CLINICAL TRIAL: NCT02448160
Title: Study Into the Effects of Albumin Replacement Therapy on Renal and Circulatory Function in Patients Implanted With the Alfapump
Brief Title: Alfapump-albumin Replacement Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-AAR-009
Record Dates: First submitted 2015-04-30; First posted 2015-05-19 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- alfapump with albumin treatment (Experimental): patients implanted with an alfapump, receiving intermittent salt-poor Human Albumin solution treatment
  Interventions: Device: alfapump; Drug: salt-poor Human Albumin solution

INTERVENTIONS:
Device: alfapump — Implantation of alfapump
  Other Names: automated low flow ascites pump
Drug: salt-poor Human Albumin solution — Patients implanted with an alfapump will receive intermittent salt-poor human albumin solution
  Other Names: Human albumin

SUMMARY:
The study will be a single centre, open-label trial. The patients will have a diagnosis of refractory ascites and will meet specified inclusion/exclusion criteria Informed consent will be obtained from all patients. All patients will have an alfapump surgically inserted and in addition will receive 8g of salt-poor Human Albumin Solution (20%) per 1 litre of Ascites drained. This Intravenous administration will be intermittent (every month) and will take place as a day patient. Patients will also receive standard of care, which may include, but is not limited to, administration of diuretics, paracentesis and consideration for orthotopic liver transplantation.

DETAILED DESCRIPTION:
The study will be a single centre, open-label trial. The patients will have a diagnosis of refractory ascites and will meet specified inclusion/exclusion criteria Informed consent will be obtained from all patients. All patients will have an alfapump surgically inserted and in addition will receive 8g of salt-poor Human Albumin Solution (20%) per 1 litre of Ascites drained. This Intravenous administration will be intermittent (every 2 weeks) and will take place as a day patient. Patients will also receive standard of care, which may include, but is not limited to, administration of diuretics, paracentesis and consideration for orthotopic liver transplantation.

The primary objective of the study is to assess whether intermittent human albumin replacement in accordance with large volume paracentesis guidelines (8g/L ascites drained) can prevent the development of renal dysfunction at the 3-month assessment. This would potentially guide the clinical use of the alfapump system.

The secondary objectives of the study are to address the objectives of a previous alfa pump study /sub study, to allow comparison of the proposed study data to that generated in the previous studies. These will be measured at the 1-month and 3-month time points.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females (determined by serum pregnancy test) ≥ 18 years of age. Women of childbearing age must be prepared to use at least 1 effective (≤1% failure rate) method of contraception during the course of the study
2. Cirrhosis of the liver defined by histological and/or clinical, and/or radiological criteria
3. Presenting with refractory ascites* and requiring periodic large volume paracentesis (large volume defined as ≥ 5 L to accord with the clinical guidance of EASL, European Association for the Study of the Liver, which recommends withdrawal of 5 L should precipitate administration of albumin).
4. Capable of giving written informed consent, willing to comply with study procedures and ability to operate the device

Exclusion Criteria:

1. Gastrointestinal haemorrhage over the last 7 days
2. Renal failure defined as serum creatinine higher than or equal to 2 mg/dl
3. Severe coagulopathy defined as prothrombin time greater than 40% more than Upper Limit of Normal
4. Platelet count of less than 40,000 / μL unless platelet therapy is given at the time of surgery
5. Clinical Evidence of recurrent bacterial peritonitis, defined as 2 or more episodes over the last 6 months or a single episode within the last 2 weeks
6. Clinical evidence of recurrent urinary infections, defined as 2 or more episodes over the last 6 months or a single episode within the last 2 weeks
7. Clinical evidence of loculated ascites
8. Advanced hepatocellular carcinoma, defined as exceeding Milan criteria
9. Obstructive uropathy, residual urinary volume exceeding 100ml, or any bladder anomaly which might contraindicate implantation of the device
10. Concurrently implanted with any other Active Implantable Medical Device, including, but not limited to cardiac pacemaker or cardiovertering defibrillator
11. Pregnant females or females anticipating pregnancy during study period
12. Patients currently enrolled in another interventional clinical study
13. Other concomitant disease or condition likely to significantly decrease life expectancy or present anaesthetic risk (e.g., moderate to severe congestive heart failure)
14. Known presence of human immunodeficiency virus (HIV)
15. Immuno-modulatory treatment (including azathioprine, methotrexate, anti-TNF therapies) used within last 4 months
16. Known or suspected hepatic or extra hepatic malignancy, unless adequately treated or in complete remission for ≥ 3 years
17. BMI>40 presenting a risk for surgery and tunnelled lines
18. Patients with contraindications for general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To assess whether intermittent human albumin replacement in accordance with large volume paracentesis guidelines (8g/L ascites drained) can prevent the development of renal dysfunction, measured by serum creatinine | 3 months
  Measured by serum creatinine.

SECONDARY OUTCOMES:
Assessment of circulatory haemodynamics, measured by non-invasive cardiac haemodynamics | 3 months
  Measured by non-invasive cardiac haemodynamics
Assessment of cirrhosis- related complications, measured by Incidence of specific cirrhosis-related complications | 3 months
  Measured by Incidence of specific cirrhosis-related complications
Assessment of the Overall Survival at 3 months, measured by survival | 3 months
  Measured by overall survival at 3 months
Assessment of impact on nutrition, measured by changes in body weight | 3 months
  Measured by changes in the nutritional status of the patient
Assessment of impact on nutrition, measured by changes in circumference of arm | 3 months
  Measured by changes in the nutritional status of the patient
Assessment of impact on nutrition, measured by changes in tricipital skinfold | 3 months
  Measured by changes in the nutritional status of the patient
Assessment of impact on nutrition, measured by changes in handgrip | 3 months
  Measured by changes in the nutritional status of the patient
Assessment of the need for large volume paracentesis, measured by the overall requirements of paracentesis | 3 months
  Measured by the overall requirement for paracentesis
Assessment of impact on Systemic Inflammatory Response, measured by CRP | 3 months
  Measured by Inflammatory markers
Assessment of impact on Systemic Inflammatory Response, measured by cytokines | 3 months
  Measured by Inflammatory markers
Assessment of impact on Systemic Inflammatory Response, measured by function of the peripheral blood mononuclear cells | 3 months
  Measured by Inflammatory markers
Assessment of levels of bacterial DNA in serum, measured by presence of bacterial DNA in blood | 3 months
  Measured by the presence of bacterial DNA in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Jalan, Professor, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided